CLINICAL TRIAL: NCT01852123
Title: High-Sensitivity Troponin in the Evaluation of Patients With Acute Coronary Syndrome: A Randomized Controlled Trial
Brief Title: High-Sensitivity Troponin in the Evaluation of Patients With Acute Coronary Syndrome
Acronym: High-STEACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); NHS Greater Glasgow and Clyde (Other); Abbott Diagnostics Division (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: High-STEACS; SP/12/10/29922 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2013-04-29; First posted 2013-05-13 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
Keywords: High-sensitivity troponin assay; Myocardial infarction; Unstable angina; Myocardial injury; Cluster randomized trial
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early implementation (Other): The high-sensitivity troponin I assay will be implemented after a 6 month validation phase
  Interventions: Device: High-sensitivity troponin I assay
- Late implementation (Other): The high-sensitivity troponin I assay will be implemented after a 12 month validation phase
  Interventions: Device: High-sensitivity troponin I assay

INTERVENTIONS:
Device: High-sensitivity troponin I assay
  Other Names: ARCHITECT STAT high-sensitive troponin I assay

SUMMARY:
In patients with chest pain the diagnosis of a heart attack (myocardial infarction) is made where there is evidence of heart muscle damage using a blood test to measure the heart muscle protein troponin. A new a more sensitive troponin test may help us to identify patients with myocardial infarction more easily.

The investigators propose to evaluate whether use of a novel high-sensitivity troponin test to lower the threshold for diagnosis of myocardial infarction is appropriate. If increased sensitivity does not reduce specificity for the diagnosis, then this new test will improve patient outcome through better targeting of therapies for coronary heart disease. However, if increased sensitivity leads to poor specificity, then patients may be misdiagnosed and given inappropriate cardiac medications with potentially detrimental outcomes.

In ten secondary and tertiary care hospitals across Scotland, the investigators will undertake a stepped wedge cluster randomized controlled trial of the implementation of a novel high-sensitivity troponin test. The primary end-point will be the one-year rate of cardiovascular death or recurrent myocardial infarction. This will establish whether the introduction of this high-sensitivity troponin test into routine clinical practice is beneficial to patient management and outcomes.

A subset of patients will be asked to give consent for inclusion into a sub-study that will permit storage of blood samples and will require the completion of a survey during the index admission and after 6 and 12 months of follow up.

ELIGIBILITY:
Inclusion criteria:

* Suspected acute coronary syndrome
* Troponin I measurement as part of routine clinical care

Exclusion criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48282 (Actual)
Dates: Start 2013-06-10 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Recurrent myocardial infarction or cardiovascular death at 1 year | 1 year

SECONDARY OUTCOMES:
Duration of stay | Initial episode
  Duration of the index hospital stay, an expected average of 2 weeks
Recurrent myocardial infarction | 1 year
Unplanned coronary revascularization | 1 year
Cardiovascular death | 1 year
All cause death | 1 year
Heart failure hospitalization | 1 year
Major hemorrhage | 1 year
Minor hemorrhage | 1 year
Recurrent unplanned hospitalization excluding acute coronary syndrome | 30 days
Non-cardiovascular death | 1 year

OTHER OUTCOMES:
Physician diagnosis on discharge | Duration of the index hospital stay, an expected average of 2 weeks
Sensitivity and specificity of sex-specific thresholds for the diagnosis of myocardial infarction | 3 months
Evaluate thresholds to rule out myocardial infarction on presentation and change criteria to rule in myocardial infarction with serial sampling. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas L Mills, MD, PhD, Principal Investigator — University of Edinburgh; Ian Ford, PhD, Study Chair — University of Glasgow
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Lothian, United Kingdom

REFERENCES:
- [Result] Shah AS, Anand A, Sandoval Y, Lee KK, Smith SW, Adamson PD, Chapman AR, Langdon T, Sandeman D, Vaswani A, Strachan FE, Ferry A, Stirzaker AG, Reid A, Gray AJ, Collinson PO, McAllister DA, Apple FS, Newby DE, Mills NL; High-STEACS investigators. High-sensitivity cardiac troponin I at presentation in patients with suspected acute coronary syndrome: a cohort study. Lancet. 2015 Dec 19;386(10012):2481-8. doi: 10.1016/S0140-6736(15)00391-8. Epub 2015 Oct 8. PMID 26454362
- [Derived] Lee KK, Doudesis D, Ferry AV, Chapman AR, Kimenai DM, Fujisawa T, Bularga A, Lowry MTH, Taggart C, Schulberg S, Wereski R, Tuck C, Strachan FE, Newby DE, Anand A, Shah ASV, Mills NL; High-STEACS Investigators. Implementation of a high sensitivity cardiac troponin I assay and risk of myocardial infarction or death at five years: observational analysis of a stepped wedge, cluster randomised controlled trial. BMJ. 2023 Nov 27;383:e075009. doi: 10.1136/bmj-2023-075009. PMID 38011922
- [Derived] Lowry MTH, Doudesis D, Boeddinghaus J, Kimenai DM, Bularga A, Taggart C, Wereski R, Ferry AV, Stewart SD, Tuck C, Koechlin L, Nestelberger T, Lopez-Ayala P, Hure G, Lee KK, Chapman AR, Newby DE, Anand A, Collinson PO, Mueller C, Mills NL; High-STEACS Investigators. Troponin in early presenters to rule out myocardial infarction. Eur Heart J. 2023 Aug 7;44(30):2846-2858. doi: 10.1093/eurheartj/ehad376. PMID 37350492
- [Derived] Neumann JT, Twerenbold R, Ojeda F, Aldous SJ, Allen BR, Apple FS, Babel H, Christenson RH, Cullen L, Di Carluccio E, Doudesis D, Ekelund U, Giannitsis E, Greenslade J, Inoue K, Jernberg T, Kavsak P, Keller T, Lee KK, Lindahl B, Lorenz T, Mahler SA, Mills NL, Mokhtari A, Parsonage W, Pickering JW, Pemberton CJ, Reich C, Richards AM, Sandoval Y, Than MP, Toprak B, Troughton RW, Worster A, Zeller T, Ziegler A, Blankenberg S; ARTEMIS study group. Personalized diagnosis in suspected myocardial infarction. Clin Res Cardiol. 2023 Sep;112(9):1288-1301. doi: 10.1007/s00392-023-02206-3. Epub 2023 May 2. PMID 37131096
- [Derived] Taggart C, Monterrubio-Gomez K, Roos A, Boeddinghaus J, Kimenai DM, Kadesjo E, Bularga A, Wereski R, Ferry A, Lowry M, Anand A, Lee KK, Doudesis D, Manolopoulou I, Nestelberger T, Koechlin L, Lopez-Ayala P, Mueller C, Mills NL, Vallejos CA, Chapman AR. Improving Risk Stratification for Patients With Type 2 Myocardial Infarction. J Am Coll Cardiol. 2023 Jan 17;81(2):156-168. doi: 10.1016/j.jacc.2022.10.025. PMID 36631210
- [Derived] Bularga A, Taggart C, Mendusic F, Kimenai DM, Wereski R, Lowry MTH, Lee KK, Ferry AV, Stewart SS, McAllister DA, Shah ASV, Anand A, Newby DE, Mills NL, Chapman AR; High-Sensitivity Troponin in the Evaluation of Patients with Suspected Acute Coronary Syndrome (High-STEACS) Investigators. Assessment of Oxygen Supply-Demand Imbalance and Outcomes Among Patients With Type 2 Myocardial Infarction: A Secondary Analysis of the High-STEACS Cluster Randomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2220162. doi: 10.1001/jamanetworkopen.2022.20162. PMID 35816305
- [Derived] Doudesis D, Lee KK, Yang J, Wereski R, Shah ASV, Tsanas A, Anand A, Pickering JW, Than MP, Mills NL; High-STEACS Investigators. Validation of the myocardial-ischaemic-injury-index machine learning algorithm to guide the diagnosis of myocardial infarction in a heterogenous population: a prespecified exploratory analysis. Lancet Digit Health. 2022 May;4(5):e300-e308. doi: 10.1016/S2589-7500(22)00025-5. PMID 35461689
- [Derived] Wereski R, Kimenai DM, Taggart C, Doudesis D, Lee KK, Lowry MTH, Bularga A, Lowe DJ, Fujisawa T, Apple FS, Collinson PO, Anand A, Chapman AR, Mills NL. Cardiac Troponin Thresholds and Kinetics to Differentiate Myocardial Injury and Myocardial Infarction. Circulation. 2021 Aug 17;144(7):528-538. doi: 10.1161/CIRCULATIONAHA.121.054302. Epub 2021 Jun 25. PMID 34167318
- [Derived] Hung J, Roos A, Kadesjo E, McAllister DA, Kimenai DM, Shah ASV, Anand A, Strachan FE, Fox KAA, Mills NL, Chapman AR, Holzmann MJ. Performance of the GRACE 2.0 score in patients with type 1 and type 2 myocardial infarction. Eur Heart J. 2021 Jul 8;42(26):2552-2561. doi: 10.1093/eurheartj/ehaa375. PMID 32516805
- [Derived] Lee KK, Ferry AV, Anand A, Strachan FE, Chapman AR, Kimenai DM, Meex SJR, Berry C, Findlay I, Reid A, Cruickshank A, Gray A, Collinson PO, Apple FS, McAllister DA, Maguire D, Fox KAA, Newby DE, Tuck C, Keerie C, Weir CJ, Shah ASV, Mills NL; High-STEACS Investigators. Sex-Specific Thresholds of High-Sensitivity Troponin in Patients With Suspected Acute Coronary Syndrome. J Am Coll Cardiol. 2019 Oct 22;74(16):2032-2043. doi: 10.1016/j.jacc.2019.07.082. PMID 31623760
- [Derived] Chapman AR, Adamson PD, Shah ASV, Anand A, Strachan FE, Ferry AV, Lee KK, Berry C, Findlay I, Cruikshank A, Reid A, Gray A, Collinson PO, Apple F, McAllister DA, Maguire D, Fox KAA, Vallejos CA, Keerie C, Weir CJ, Newby DE, Mills NL; High-STEACS Investigators. High-Sensitivity Cardiac Troponin and the Universal Definition of Myocardial Infarction. Circulation. 2020 Jan 21;141(3):161-171. doi: 10.1161/CIRCULATIONAHA.119.042960. Epub 2019 Oct 7. PMID 31587565
- [Derived] Bularga A, Lee KK, Stewart S, Ferry AV, Chapman AR, Marshall L, Strachan FE, Cruickshank A, Maguire D, Berry C, Findlay I, Shah ASV, Newby DE, Mills NL, Anand A. High-Sensitivity Troponin and the Application of Risk Stratification Thresholds in Patients With Suspected Acute Coronary Syndrome. Circulation. 2019 Nov 5;140(19):1557-1568. doi: 10.1161/CIRCULATIONAHA.119.042866. Epub 2019 Sep 1. PMID 31475856
- [Derived] Ferry AV, Anand A, Strachan FE, Mooney L, Stewart SD, Marshall L, Chapman AR, Lee KK, Jones S, Orme K, Shah ASV, Mills NL. Presenting Symptoms in Men and Women Diagnosed With Myocardial Infarction Using Sex-Specific Criteria. J Am Heart Assoc. 2019 Sep 3;8(17):e012307. doi: 10.1161/JAHA.119.012307. Epub 2019 Aug 20. PMID 31431112
- [Derived] Neumann JT, Twerenbold R, Ojeda F, Sorensen NA, Chapman AR, Shah ASV, Anand A, Boeddinghaus J, Nestelberger T, Badertscher P, Mokhtari A, Pickering JW, Troughton RW, Greenslade J, Parsonage W, Mueller-Hennessen M, Gori T, Jernberg T, Morris N, Liebetrau C, Hamm C, Katus HA, Munzel T, Landmesser U, Salomaa V, Iacoviello L, Ferrario MM, Giampaoli S, Kee F, Thorand B, Peters A, Borchini R, Jorgensen T, Soderberg S, Sans S, Tunstall-Pedoe H, Kuulasmaa K, Renne T, Lackner KJ, Worster A, Body R, Ekelund U, Kavsak PA, Keller T, Lindahl B, Wild P, Giannitsis E, Than M, Cullen LA, Mills NL, Mueller C, Zeller T, Westermann D, Blankenberg S; COMPASS-MI Study Group. Application of High-Sensitivity Troponin in Suspected Myocardial Infarction. N Engl J Med. 2019 Jun 27;380(26):2529-2540. doi: 10.1056/NEJMoa1803377. PMID 31242362
- [Derived] Chapman AR, Fujisawa T, Lee KK, Andrews JP, Anand A, Sandeman D, Ferry AV, Stewart S, Marshall L, Strachan FE, Gray A, Newby DE, Shah ASV, Mills NL. Novel high-sensitivity cardiac troponin I assay in patients with suspected acute coronary syndrome. Heart. 2019 Apr;105(8):616-622. doi: 10.1136/heartjnl-2018-314093. Epub 2018 Nov 15. PMID 30442743
- [Derived] Chapman AR, Hesse K, Andrews J, Lee KK, Anand A, Shah ASV, Sandeman D, Ferry AV, Jameson J, Piya S, Stewart S, Marshall L, Strachan FE, Gray A, Newby DE, Mills NL. High-Sensitivity Cardiac Troponin I and Clinical Risk Scores in Patients With Suspected Acute Coronary Syndrome. Circulation. 2018 Oct 16;138(16):1654-1665. doi: 10.1161/CIRCULATIONAHA.118.036426. PMID 30354460
- [Derived] Shah ASV, Anand A, Strachan FE, Ferry AV, Lee KK, Chapman AR, Sandeman D, Stables CL, Adamson PD, Andrews JPM, Anwar MS, Hung J, Moss AJ, O'Brien R, Berry C, Findlay I, Walker S, Cruickshank A, Reid A, Gray A, Collinson PO, Apple FS, McAllister DA, Maguire D, Fox KAA, Newby DE, Tuck C, Harkess R, Parker RA, Keerie C, Weir CJ, Mills NL; High-STEACS Investigators. High-sensitivity troponin in the evaluation of patients with suspected acute coronary syndrome: a stepped-wedge, cluster-randomised controlled trial. Lancet. 2018 Sep 15;392(10151):919-928. doi: 10.1016/S0140-6736(18)31923-8. Epub 2018 Aug 28. PMID 30170853
- [Derived] Miller-Hodges E, Anand A, Shah ASV, Chapman AR, Gallacher P, Lee KK, Farrah T, Halbesma N, Blackmur JP, Newby DE, Mills NL, Dhaun N. High-Sensitivity Cardiac Troponin and the Risk Stratification of Patients With Renal Impairment Presenting With Suspected Acute Coronary Syndrome. Circulation. 2018 Jan 30;137(5):425-435. doi: 10.1161/CIRCULATIONAHA.117.030320. Epub 2017 Oct 4. PMID 28978551
- [Derived] Chapman AR, Anand A, Boeddinghaus J, Ferry AV, Sandeman D, Adamson PD, Andrews J, Tan S, Cheng SF, D'Souza M, Orme K, Strachan FE, Nestelberger T, Twerenbold R, Badertscher P, Reichlin T, Gray A, Shah ASV, Mueller C, Newby DE, Mills NL. Comparison of the Efficacy and Safety of Early Rule-Out Pathways for Acute Myocardial Infarction. Circulation. 2017 Apr 25;135(17):1586-1596. doi: 10.1161/CIRCULATIONAHA.116.025021. Epub 2016 Dec 29. PMID 28034899

DOCUMENTS (2):
  • Study Protocol (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT01852123/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT01852123/SAP_001.pdf